CLINICAL TRIAL: NCT02493972
Title: Interest of the Manual Exploration as a Supplement to the Coelioscopy in the Evaluation of the Resectability of Peritoneal Carcinosis
Acronym: CARPEMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00615-44
Record Dates: First submitted 2015-06-26; First posted 2015-07-10 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer With Peritoneal Carcinosis
Keywords: ovarian cancer; peritoneal carcinosis; manual exploration; surgery; GelPort
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- manual exploration by GelPort (Experimental): manual exploration in supplement of coelioscopy before laparotomy
  Interventions: Procedure: GelPort; Procedure: laparotomy

INTERVENTIONS:
Procedure: GelPort — Manual exploration of the peritoneal carcinosis by the system GelPort ® with calculation of peritoneal cancer index for evaluation of the resectability
Procedure: laparotomy — laparotomy will be performed if indication confirmed by manual exploration

SUMMARY:
This is a Multicenter prospective diagnostic study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age Patient
* Woman presenting a peritoneal carcinosis presumed ovarian origin
* Coelioscopy (1st intent or recurrence) planned or performed in the last 4 weeks for laparotomy. The peritoneal cancer index of Sugarbaker must be available.
* WHO 0 - 2
* Membership in a social security system
* Patient having given her written consent

Exclusion Criteria:

* Male
* Contraindication in the coelioscopy
* Any associated medical or psychological condition which could compromise the capacity of the patient to participate in the study
* Patient deprived of freedom, under guardianship or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
evaluate the number of patients with or without laparotomy after evaluation of the resectability by coelioscopy and coelioscopy more manual exploration | 1 month after inclusion

SECONDARY OUTCOMES:
Number of patients with complications (eventrations, infections, pains) after manual exploration | 1 month after inclusion
Number of patients with parietal metastases | 1 month after inclusion

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU, Amiens
  - Centre Françis Baclesse, Caen
  - CHU, Caen
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Henri Becquerel, Rouen